CLINICAL TRIAL: NCT03987438
Title: Diabetes Mellitus, Impaired Glucose Tolerance and Gestational Diabetes Mellitus Intervention Action-Leading Trial- Impaired Glucose Tolerance Study (DIGITAL-I Study)
Brief Title: A Behavioral Intervention to Prevent Impaired Glucose Tolerance Diabetes Mellitus (DIGITAL-I)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIGITAL-I-2019
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes
Keywords: Behavioral intervention; Imparied glucose tolerance; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral intervention (Experimental): Participants randomized to the behavioral intervention group will be provided with a mobile APP which incorporates behavioral support including health knowledge education, mental health counseling, diet advice, exercise guidance and weight management. Meanwhile, the behavioral support will be modified by endocrinologists, dieticians, sports medicine professionals and psychologists individually based on the feedback of their performance recorded in the APP. Every three months, participants in the intervention group will be back to their research centers and be collected with information including HbA1c levels, blood pressure, heart rate tests and adverse events. Investigators conduct face-to-face health education, lifestyle guidance, mobile APP software inspection. Every one year, 75g OGTT (0min,60min, 120min points of blood glucose and insulin levels), liver and kidney function, blood lipids, glycosylated hemoglobin, urine routine and electrocardiogram will be evaluated.
  Interventions: Behavioral: Lifestyle intervention with APP
- Control group (No Intervention): Participants randomized to the control group have regular care in their local hospitals. Every three months, participants in the intervention group will be back to their research centers and be collected with information including HbA1c levels, blood pressure, heart rate tests and adverse events. Every one year, 75g OGTT (0min,60min, 120min points of blood glucose and insulin levels), liver and kidney function, blood lipids, glycosylated hemoglobin, urine routine and electrocardiogram will be evaluated.

INTERVENTIONS:
Behavioral: Lifestyle intervention with APP — The lifestyle intervention will be launched by an APP installed in participants' private mobile phones, including health knowledge education, mental health counseling, smart diet advice, intelligent exercise guidance, and target weight management. Nutrition recommendation is conducted according to the Chinese Dietary Guide, Chinese and International Guidelines of Gestation Diabetes Management. Exercise guidance is given based on the Guidelines for National Fitness of China, Chinese and International Guidelines of Gestation Diabetes Management. Psychological support is given by sending education articles on mental health. Participants are encouraged to update data about their diet, exercise and body weight through the APP. The face to face education class will be conducted by an obstetrician, an endocrinologist and a nutritionist together to modify the behavioral supports individually based on the feedback of their characteristics and performance recorded in the APP.
  Arms: Behavioral intervention

SUMMARY:
The national epidemiological survey showed that the prevalence rate of pre-diabetes was up to 35.7% in China. Previous study indicated that lifestyle intervention in people with impaired glucose tolerance could delay the onset of type 2 diabetes. However, patients with pre-diabetes do not pay enough attention to their glucose metabolism, and most of them rarely monitor their blood glucose. With the increasing use of smartphones, mobile applications (APPs) can be applied in the education and management of chronic diseases, including diabetes. Thus, the investigators will conduct a multi-centered, two-armed, open-labeled, randomized controlled trial to evaluate whether the behavioral intervention by a mobile APP can prevent the occurrence of diabetes in people with impaired glucose tolerance.

The investigators hypothesize that behavioral intervention in pre-diabetes with using a mobile APP that incorporates nutrition, exercise and psychological support from trained professional doctors will:

1. Reduce the risk of the onset of diabetes in people with impaired glucose tolerance.
2. Increase the reversal rate of becoming normal glucose tolerance and reduce the levels of glycosylated hemoglobin in pre-diabetes.

DETAILED DESCRIPTION:
Participants from fourteen research centers in the mainland of China will be recruited in the study. People will be screened for a 75g oral glucose tolerance test (OGTT). The patients whose fasting glucose between 6.1mmol/L and 7.0mmol/L or 2-hour value between 7.8mmol/L and 11.1mmol/L will be diagnosed with impaired glucose tolerance and recommended to participate in the study.

People who meet the eligibility criteria and who are willing to provide informed consent will be enrolled and randomized to behavioral intervention group and control group. People in the behavioral intervention group will be educated and monitored by a mobile APP that provides behavioral support including health knowledge education, mental health counseling, smart diet advice, intelligent exercise guidance, and target weight management. Meanwhile, the behavioral support will be modified by endocrinologists, dieticians, sports medicine professionals and psychologists individually based on the feedback of their characteristics and performance recorded in the APP. Participants randomized to the control group only have regular care in their local hospitals.

Every three months, participants in the intervention group will be back to their research centers and be collected with information including HbA1c levels, blood pressure, heart rate tests, adverse events, combined medications and health checklists. Investigators conduct face-to-face health education, lifestyle guidance and mobile APP software inspection. Every one year, 75g OGTT (0min, 60min, 120min points of blood glucose and insulin levels), liver and kidney function, blood lipids, glycosylated hemoglobin, urine routine and electrocardiogram will be evaluated in both of the group. Investigators will compare the diabetes risk in the two groups to evaluate whether behavioral intervention with a mobile APP can reduce the risk of the onset of diabetes in people with impaired glucose tolerance. Investigators also will compare the reversal rate of becoming normal glucose tolerance in prediabetes and the changes of glycosylated hemoglobin levels in both groups. Behavioral intervention with the APP will last for two years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Impaired glucose tolerance will be diagnosed by a 75g OGTT according to the criteria of World Health Organization as a fasting plasma glucose level between 6.1 mmol/L and 7.0 mmol/L, or 2-hour value between 7.8 mmol/L and 11.1 mmol/L
* Willing to keep reading the education articles and supporting materials that delivered by the mobile APP
* Willing to provide informed consent

Exclusion Criteria:

* Pregnant women, pregnant or lactating women (Can be reassessed after childbirth or after breastfeeding)
* Inconvenient to move, far away from the center to limit follow-up, more than 2 hours drive from the center
* Cannot complete the test because of planning migration
* Schizophrenia, manic depression, drug or alcohol addicts
* Cancer patients who have been treated in the past 5 years
* HIV positive (report)
* Active tuberculosis
* Patients with severe CVD (Myocardial infarction, heart failure, stroke) or pulmonary embolism in the past 6 months
* Unstable angina or resting angina; history of cardiac arrest; severe arrhythmia; uncontrolled atrial fibrillation (heart rate not less than 100 beats / min); cardiac function by New York Cardiology Society Grade III ~ IV; acute myocarditis, pericarditis or hypertrophic cardiomyopathy; clinically significant aortic stenosis; severe left bundle branch block or installation of a pacemaker (unless agreed by a cardiologist); history of defibrillation; aortic aneurysm diameter > 7cm or history of aortic rupture; history of heart transplantation; resting heart rate <45 beats / min or > 100 beats / min
* Cirrhosis; Cushing's syndrome; acromegaly; long-term application of glucocorticoids
* Serum creatinine is 2 times higher than the upper limit of normal; currently undergoing dialysis
* Chronic anoxia diseases such as emphysema, pulmonary heart disease, etc.
* Rheumatic heart disease; congenital heart disease
* Organ transplantation patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1336 (Estimated)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The risk of diabetes mellitus (DM) in patients with impaired glucose tolerance | 2 years
  DM will be diagnosed by a 75g OGTT according to the World Health Organization criteria as fasting plasma glucose level 7.0 mmol/L or more, or 2-hour value 11.1 mmol/L or more. Investigators will compare the diabetes risk in the two groups to evaluate whether behavioral intervention with a mobile APP can reduce the risk of the onset of diabetes in people with impaired glucose tolerance.

SECONDARY OUTCOMES:
Reversal rate of becoming normal glucose tolerance in pre-diabetes | 2 years
  Every one year, 75g OGTT (0min,60min, 120min points of blood glucose and insulin levels) will be evaluated in both of the group. Investigators will compare the reversal rate of becoming normal glucose tolerance in pre-diabetes.
Changes in glycosylated hemoglobin levels. | 2 years
  Glycosylated hemoglobin levels will be recorded at the beginning, middle and end of the study. Investigators will compare the changes in glycosylated hemoglobin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tianpei Hong, MD,PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital YanQing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No